CLINICAL TRIAL: NCT04404933
Title: An Observational Study of Diagnostic Criteria, Clinical Features and Management of Opioid-induced Constipation (OIC) in Patients With Cancer Pain
Brief Title: Study of Opioid-Induced Constipation 2 Project
Acronym: StOIC-2
Status: Completed | Type: Observational
Sponsor: Royal Surrey County Hospital NHS Foundation Trust (Other)
Collaborators: Kyowa Hakko Kirin UK, Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: StOIC-2 Project
Record Dates: First submitted 2020-05-22; First posted 2020-05-28 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-04

CONDITIONS: Opioid-induced Constipation; Cancer; Cancer Pain
Keywords: Opioid-induced constipation
MeSH Terms: conditions — Opioid-Induced Constipation; Neoplasms; Cancer Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Treatment algorithm for OIC — Treatment Algorithm for OIC

SUMMARY:
The aim of the project is to investigate OIC in a real world / diverse group of patients with cancer.

The objectives of the project are to determine: a) efficacy of a treatment algorithm to manage OIC; b) efficacy of conventional laxatives to manage OIC; c) efficacy of PAMORAs / other interventions to manage OIC.

DETAILED DESCRIPTION:
StOIC-2 is an observational study of routine clinical practice, and will involve four assessments over a period of 28 days (3 face to face; 1 telephone). Participants for StOIC 2 study will be identified from StOIC 1 study (CancerTrials.gov registry reference number - NCT04350112). Visit 1 for StOIC 2 study will correspond to the assessment for StOIC 1 study.

Patients will be managed according to a treatment algorithm (see below), which is based on a review of the evidence (and which is the basis of the Multinational Association for Supportive Care in Cancer (MASCC) guideline on the treatment of constipation in patients with advanced cancer). The decision to change treatment is based on efficacy / lack of efficacy (as determined by the Bowel Function Index (see below), or the development of adverse effects.

Step 1: Conventional Laxatives

* Choice of laxatives at the discretion of the clinical team
* Combination of softener and stimulant laxative
* Laxatives to be prescribed on a regular basis

Step 2: Peripherally acting mu opioid receptor antagonist (PAMORA)

* Choice of PAMORA at the discretion of clinical team
* Either oral naloxegol or subcutaneous methylnaltrexone
* PAMORA to be prescribed on a regular basis

Step 3: PAMORA + Conventional Laxatives

* Choice of combination at the discretion of the PI/clinical team
* Combination to be prescribed on a regular basis

Step 4: Other options

- Choice of other option at discretion of clinical team:

* Bowel cleansing preparations (e.g. Picolax)
* Suppositories
* Enemas
* Manual evacuation
* Other drugs (e.g. lubiprostone, prucalopride)

The following data will be collected: a) demographic data - age, gender, ethnicity; b) cancer diagnosis; c) opioid medications - drug, formulation, dose; d) laxative medications - drug, formulation, dose (every visit); e) Eastern Cooperative Oncology Group performance status.

The participants will also be asked to complete;

1. Bowel Function Index (BFI) - every visit. The BFI is a validated, 3 item, patient reported tool for assessing the treatment of OIC. A BFI score of > 30 indicates suboptimally treated OIC.
2. Patient Assessment of Constipation - Quality of Life Questionnaire (PAC-QOL) - first and last visit. The PAC-QOL is a validated, 28 item, patient reported tool for assessing the impact of constipation over time.
3. Memorial Symptom Assessment Scale - Short Form (MSAS-SF) - first and last visit. The MSAS-SF is a validated, 32 item, patient reported tool for assessing physical and psychological symptoms in cancer patients.

Data will also be collected on adverse effects from medication / interventions, and reasons for withdrawal from the study.

ELIGIBILITY:
Inclusion Criteria:

* As per StOIC 1: age > 18yr; diagnosis of cancer; diagnosis of cancer pain; receipt of regular opioids for at least one week
* Diagnosis of OIC as defined by the Rome IV criteria (Lacy et al, 2016)
* Diagnosis of inadequately treated OIC as defined by BFI > 30

Exclusion Criteria:

* As per StOIC 1: inability to give informed consent; inability yo complete questionnaire
* Prognosis > 1 month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants may be inpatients, outpatients, day centre patients and home care patients at the sites conducting the research
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Resolution of OIC | 28 days
  BFI < 30

SECONDARY OUTCOMES:
Improvement in BFI | 28 days
  BFI improved by 12

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Davies, MD, Principal Investigator — Consultant Palliative Medicine
Locations (16):
- United Kingdom (16):
  - Royal Cornwall Hospital, Truro, Cornwall
  - Brighton & Sussex University Hospitals, Brighton, East Sussex
  - Leckhampton Court Hospice, Cheltenham, Gloucestershire
  - Hospice of St. Francis, Berkhamstead, Hertfordshire
  - Heart of Kent Hospice, Maidstone, Kent
  - Wisdom Hospice, Rochester, Kent
  - St. Raphael's Hospice, Cheam, London
  - Nottingham University Hospitals, Nottingham, Nottinghamshire
  - St Margaret's Hospice, Yeovil, Somerset
  - St. Giles Hospice, Lichfield, Staffordshire
  - Royal Surrey County Hospital, Guildford, Surrey
  - Birmingham St. Mary's Hospice, Birmingham, West Midlands
  - St. Catherine's Hospice, Crawley, West Sussex
  - St. Gemma's Hospice, Leeds, Yorkshire
  - Wheatfields Hospice, Leeds, Yorkshire
  - St. Luke's Hospice, Sheffield, Yorkshire

IPD SHARING:
Plan to Share IPD: No
Currently, there are no plans to make IPD available to other researchers

REFERENCES:
- [Result] Davies A, Leach C, Caponero R, Dickman A, Fuchs D, Paice J, Emmanuel A. MASCC recommendations on the management of constipation in patients with advanced cancer. Support Care Cancer. 2020 Jan;28(1):23-33. doi: 10.1007/s00520-019-05016-4. Epub 2019 Aug 9. PMID 31396746
- [Result] Rentz AM, Yu R, Muller-Lissner S, Leyendecker P. Validation of the Bowel Function Index to detect clinically meaningful changes in opioid-induced constipation. J Med Econ. 2009;12(4):371-83. doi: 10.3111/13696990903430481. PMID 19912069
- [Result] Argoff CE, Brennan MJ, Camilleri M, Davies A, Fudin J, Galluzzi KE, Gudin J, Lembo A, Stanos SP, Webster LR. Consensus Recommendations on Initiating Prescription Therapies for Opioid-Induced Constipation. Pain Med. 2015 Dec;16(12):2324-37. doi: 10.1111/pme.12937. Epub 2015 Nov 19. PMID 26582720
- [Result] Marquis P, De La Loge C, Dubois D, McDermott A, Chassany O. Development and validation of the Patient Assessment of Constipation Quality of Life questionnaire. Scand J Gastroenterol. 2005 May;40(5):540-51. doi: 10.1080/00365520510012208. PMID 16036506
- [Result] Chang VT, Hwang SS, Feuerman M, Kasimis BS, Thaler HT. The memorial symptom assessment scale short form (MSAS-SF). Cancer. 2000 Sep 1;89(5):1162-71. doi: 10.1002/1097-0142(20000901)89:53.0.co;2-y. PMID 10964347
- [Derived] Davies AN, Leach C, Butler C, Patel SD, Shorthose K, Batsari K. Opioid-induced constipation: a stepwise treatment algorithm feasibility study. BMJ Support Palliat Care. 2023 Dec 7;13(e2):e446-e453. doi: 10.1136/bmjspcare-2020-002754. PMID 34348942